CLINICAL TRIAL: NCT03983720
Title: Can Fatigability Neuromuscular Explain Chronic Fatigue in People With Multiple Sclerosis?
Acronym: FatSEP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low inclusion rates
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 19CH030; 2019-A00427-50 (Other: ID-RCB)
Record Dates: First submitted 2019-06-07; First posted 2019-06-12 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Sclerosis, Multiple
Keywords: Sleep assessment; Neuromuscular Fatigability; Multiple sclerosis; Chronic fatigue
MeSH Terms: conditions — Multiple Sclerosis | interventions — Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patient with multiple sclerosis and lowly fatigued (Experimental): Patient with multiple sclerosis and lowly fatigued will be included.
  They will have:
  Visit 1 (day 0) = Questionnaires, blood sample, cardiopulmonary evaluation, capacity of muscular oxygen extraction, sleep assessment Visit 2 (day 15) = Neuromuscular evaluation Visit 3 (day 30) = Metabolic fatigue
  Interventions: Other: Evaluation of degree chronic fatigue.; Other: Questionnaires; Biological: Blood sample; Other: Cardiopulmonary evaluation; Device: Capacity of muscular oxygen extraction; Device: Sleep assessment; Device: Metabolic fatigue; Other: Neuromuscular evaluation
- Patient with multiple sclerosis and highly fatigued (Experimental): Patient with multiple sclerosis and highly fatigued will be included. They will have:
  Visit 1 (day 0) = Questionnaires, blood sample, cardiopulmonary evaluation, capacity of muscular oxygen extraction, sleep assessment Visit 2 (day 15) = Neuromuscular evaluation Visit 3 (day 30) = Metabolic fatigue
  Interventions: Other: Evaluation of degree chronic fatigue.; Other: Questionnaires; Biological: Blood sample; Other: Cardiopulmonary evaluation; Device: Capacity of muscular oxygen extraction; Device: Sleep assessment; Device: Metabolic fatigue; Other: Neuromuscular evaluation
- Healthy subjects (Active Comparator): Healthy subjects will be included. They will have:
  Visit 1 (day 0) = Questionnaires, blood sample, cardiopulmonary evaluation, capacity of muscular oxygen extraction, sleep assessment Visit 2 (day 15) = Neuromuscular evaluation Visit 3 (day 30) = Metabolic fatigue
  Interventions: Other: Questionnaires; Biological: Blood sample; Other: Cardiopulmonary evaluation; Device: Capacity of muscular oxygen extraction; Device: Sleep assessment; Device: Metabolic fatigue; Other: Neuromuscular evaluation

INTERVENTIONS:
Other: Evaluation of degree chronic fatigue. — Evaluation of degree chronic fatigue with the results of survey Fatigue Severity Scale (FSS) and Modified Fatigue Impact Scale (MFIS). This result will allow to divide patients in groups : lowly fatigued and highly fatigued.
  Arms: Patient with multiple sclerosis and highly fatigued; Patient with multiple sclerosis and lowly fatigued
Other: Questionnaires — * Fatigue Severity Scale (FSS)
  * Modified Fatigue Impact Scale (MFIS)
  * Godin Leisure-Time Exercise Questionnaire (GLTEQ)
  * Scale of life quality of multiple sclerosis (SEP-59)
  * Center for Epidemiologic Studies Depression (CES-D)
  * Pittsburgh Sleep Quality Index (PSQ-I)
Biological: Blood sample — Blood sample will be realized to evaluate anemia and inflammations.
Other: Cardiopulmonary evaluation — Cardiopulmonary evaluation will be realized with a cycle ergometer.
Device: Capacity of muscular oxygen extraction — Measure the capacity of muscular oxygen extraction with a cycle ergometer.
Device: Sleep assessment — Sleep assessment will be measured by actigraphy during 15 days.
Device: Metabolic fatigue — Metabolic fatigue will be measured by Magnetic Resonance Imaging (MRI).
Other: Neuromuscular evaluation — Neuromuscular evaluation will be measured by the composite of the results of:
  * Fatigue test
  * Measure of voluntary isometric force
  * Surface electromyography
  * Peripheral nerve stimulation
  * Transcranial Magnetic Stimulation (TMS)
  * Perceived fatigue
  * Cognitive fatigue
  * Thermoregulation

SUMMARY:
Chronic fatigue is the most common and debilitating symptom in multiple sclerosis patients. This chronic fatigue affects their quality of life by decreasing their capacity to perform simple tasks of daily life.

The aim of the present project is to determine whether deteriorated neuromuscular function (i.e. increased fatigability) is involved in this feeling of chronic fatigue. Because the causes of this feeling are multi-dimensional, a large battery of tests will allow us to better understand the origin of chronic fatigue. A better knowledge of chronic fatigue etiology will allow to optimize rehabilitation treatments to decrease the apparition/persistence of chronic fatigue and in fine improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

For Patients:

* Aged ≥ 18 and ≤ 70 years
* Men or women
* With multiple sclerosis since 2 and 25 years
* Affiliates or beneficiaries of social security scheme
* Signed consent

For Healthy volunteers:

* Aged ≥ 18 and ≤ 70 years
* Men or women
* Matched in accordance with age, sex and level of physical activity

Exclusion Criteria:

For Patients and Healthy volunteers:

* High heart rate resting
* Blood pressure > 144/94 mmHg
* Recent adjustment of drug or drug can have an impact on fatigue or stimulant for fatigue
* Taking neuroactive substances that can alter corticospinal excitability
* Contraindication at application magnetic field
* Contraindication at Magnetic Resonance Imaging (MRI)
* Currently participating in a structured exercise program
* Pregnant

For Patients only:

* Spasticity or cerebellar ataxia
* Abnormal range of motion (toe and/or ankle)
* Musculoskeletal injuries that impedes pedaling
* Appearance of symptoms of multiple sclerosis in the 90 days preceding the study

For Healthy volunteers:

- Neurological diseases, cardiovascular, musculoskeletal

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Voluntary maximum contraction | Day : 30
  Comparison the percentage of decrease in voluntary maximum contraction reported after the fatiguing task. Measured by an instrumented measuring pedal (PowerForce pedal, Model PF1.0.0.0, Radlabor GmbH, Freiburg, Germany)

SECONDARY OUTCOMES:
Neuromuscular function during the dynamic strenuous exercise | Day : 30
  Cortical activity by transcranial magnetic stimulation, evaluated by recording of the evoked motor potentials
  .
Muscle oxygen extraction capacity | Day : 30
  Measured by near-infrared spectroscopy (NIRS)
Anemia | Day : 30
  Measured by blood count in blood sample
Inflammation | Day : 30
  Measured by C-reactiv protein in blood sample
VO2 max | Day : 30
  Measured by effort test
Heart rate | Day : 30
  Measured by heart rate monitor
Cognitive fatigue | Day : 30
  Measured by Symbol Digit Modalities Test
Perceived fatigue | Day : 30
  Measured by Borg scale
Thermoregulation | Day : 30
  Measured by digestible thermometric pill (e-celcius Performance)
Sleep quality | Day : 30
  Measured by actigraphy
Muscle volume | Day : 30
  Measured by Magnetic Resonance Imaging
Metabolic fatigue | Day : 30
  Measured by a Phosphorus 31 Nuclear Magnetic Resonance test

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe CAMDESSANCHE, MD PhD, Principal Investigator — CHU DE SAINT ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No